CLINICAL TRIAL: NCT01917071
Title: The Effect of Directional Specific Thoracic Spine Mobilization on Cervial Spine Pain.
Brief Title: The Effect of Directional Specific Thoracic Spine Mobilization on Cervical Spine Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chatham University (Other)
Responsible Party: Principal Investigator, Steve Karas, Assistant Professor, Chatham University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Karasmatched
Record Dates: First submitted 2013-08-02; First posted 2013-08-06 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2013-08

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Matched Group (Experimental): Receives thoracic spine manipulation in the direction of motion limitation.
  Interventions: Other: thoracic spine manipulation

INTERVENTIONS:
Other: thoracic spine manipulation — a manual technique applied to the mid back to promote motion

SUMMARY:
Hypothesis: There is no difference in directional specific manipulation of the thoracic spine for patients with neck pain.

Patients seeking physical therapy for neck pain routinely have their thoracic spine manipulated. This study seeks to determine if directional limitations in the spine can be specifically determined and treated to decrease neck pain.

DETAILED DESCRIPTION:
Manipulation of the thoracic spine is the most commonly used manual therapy intervention by manual therapists. It is not known whether we can accurately assess and treat directional limitations in the thoracic spine to improve neck pain.

One way is to assess where the limitation is and treat it. Another method is to distract the joint. We want to know if matching the limitation to the manipulation method will give patients with neck pain better results.

The patient lays on their back. The therapist places a hand on the inferior vertebrae of the motion segment. The patient relaxes and the therapist pushes in an anterior to posterior direction either moving the vertebrae into flexion or entension.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Neck Pain; ages 18 - 60

Exclusion Criteria:

* red flags: leg weakness, night pain, history of cancer, upper motor neuron signs, infection, tumors, osteoporosis, fracture (Boissonnault, 2011) (Cleland, 2004) history of whiplash within 6 weeks, cervical stenosis, CNS involvement, signs consistent with nerve root compression, previous surgery, pending legal action

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | 2 weeks
  Objective, valid, reliable measure of function in patients with neck pain. Completed as a survey.

SECONDARY OUTCOMES:
Neck Pain | 2 weeks
  Selection of 0 to 10 level of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Steve A Karas, DSc, PT, Study Director — Chatham University
Locations (1):
- Chatham University, Pittsburgh, Pennsylvania, United States